CLINICAL TRIAL: NCT06094595
Title: Adaptation and Validation of the Logopaedic Assessment Protocol Mealtime Assessment Scale (MAS) in Paediatric Patients
Brief Title: Mealtime Assessment Scale-p Adaptation and Validation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Don Carlo Gnocchi ONLUS - Centro Bignamini, Falconara Marittima (Unknown); Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Giovanna Cristella, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: MAS-p
Record Dates: First submitted 2023-09-05; First posted 2023-10-23 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Dysphagia
Keywords: Pediatric population; Dysphagia assessment
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MAS-p administration — Each patient will be assessed the first time at mealtime by two experienced speech therapists, and scores obtained on the MAS-p will be recorded independently and blinded to each other. The two scales selected for comparison will also be administered at the same time. The assessment with the MAS-p scale will be repeated 48 hours apart, a time considered optimal in order to avoid possible bias related to the clinical improvement of the patient undergoing rehabilitation treatment, by one of the two speech therapists.

SUMMARY:
The study aims to adapt the Mealtime Assessment Scale (MAS) in a pediatric population in order to provide an observational tool compiled by swallowing professionals, in Italian, for the assessment of swallowing efficacy and safety during mealtime in an ecological setting, as mealtime administration occurs independently or by the caregiver.

DETAILED DESCRIPTION:
The study is developed in 3 phases, replicating the validation process of the original version of the MAS scale validated on the adult population, based on the studies of Hansen et al.

1 Phase - adaptation of the scale to its use in pediatric settings. The first part of the study will be aimed at performing an adaptation of the original version of the MAS scale to the pediatric population by a multidisciplinary team consisting of physicians specializing in Physical Medicine and Rehabilitation, speech pathologists, and clinical psychologists.

The MAS consists of an initial section devoted to the collection of biographical and anamnestic data. It is then divided into four subscales: 1. Structures, functions and activities that influence eating, 2. Environmental factors that influence eating, 3. Safety of swallowing during eating, 4. Efficacy of swallowing during eating, for a total of 26 items. The score of each item is calculated from 0 (normal) to 3 (severely impaired).

The scale includes a section for calculating the score and a final supplementary section without scoring concerning the need for patient compensation and cues, which is intended to provide qualitative, not quantitative, descriptive information.

It is possible to calculate a partial score obtained at the subscales concerning Safety and Swallowing Effectiveness given by the sum of the scores at the relevant items, which can be expressed as a percentage value, to facilitate quantification of the level of impairment in these aspects. The higher the score or percentage, the lower the safety and effectiveness of swallowing during the meal. The time of intake of the same is also specified.

This study aims to maintain this structure and scoring system also in adapting the scale for the pediatric population (MAS-p).

Some items will be added, modified or removed according to the physiological characteristics of the pediatric subject, in particular it is deemed necessary to include an item exploring teething with its different characteristics according to life periods, an item for sucking if it is still present. Items will be removed if they are not applicable or not explorable in the test population, such as short-term memory. An initial review of the modified scale will be discussed by the multidisciplinary team in order to assess the comprehensibility of the proposed items.

Phase 2 - preliminary study At the end of the scale modification and adaptation process, a preliminary study of the psychometric properties of the pediatric version of the scale will be carried out through a pilot study in order to confirm the validity of the structure of the new scale, to study its internal consistency, intra- and inter-rater reliability, and finally the discrimination index.

A sample of 40 subjects was identified for the validation pilot study, aged between 24 months and 18 years, recruited on an outpatient and inpatient basis from paediatric rehabilitation department of the Don Carlo Gnocchi Foundation in Florence, Meyer Hospital in Florence, Don Carlo Gnocchi Foundation in Falconara.

Each recruited patient will be observed during the consumption of an entire meal by an experienced speech therapist informed of the protocol, in the presence of the caregiver. If the patient is not suitable due to age or pathology to perform this task independently, the administration of the meal will be entrusted to the caregiver, in an attempt to observe the patient in as ecological a setting as possible, as much superimposed on the context of family life in which the meal takes place daily. For this purpose, it will also be proposed to the patient to feed himself, in addition to the personal utensils used at home, with foods of his liking, usually included in his own diet.

The duration of administration of the scale, by the speech therapist assigned to the role of observer, will depend on the time it takes the test subject to eat a meal (on average between 30 and 45 minutes). Finally, it will take 4 to 5 minutes to complete the scoring section.

For the first 10 of the 40 patients recruited, observation will be conducted by two independent operators, experts in the protocol, who will fill out the scale blind to each other in order to test inter-operator reliability.

Intra-operator reliability will be studied by administration by the same operator to the subject 48 hours after the first assessment, in order to limit possible bias due to a change in the patient's clinical condition.

A second review of the scale by the multidisciplinary team, previously described, will therefore be carried out in order to discuss and possibly further modify the items that make up the scale.

Phase 3 - validation of the MAS-p scale. This phase aims to validate the pediatric version of the MAS scale on a larger group of patients.

A sample of 200 subjects has been identified, based on the studies of Hansen et al. and the validation study of the original version of the MAS scale. The recruited subjects will be divided into groups as follows.

Group 1: sample of 100 subjects not at risk for swallowing disorders as a control group.

Group 2: sample of 100 subjects at risk of swallowing disorders, with different underlying pathology, who tolerate full or partial oral meal intake.

Group 3: 36 patients with suspected dysphagia, selected in Group 2, for whom dietary modification is expected during the period of hospitalization.

During the meal, the evaluator may talk to the patient, encourage the patient to complete the meal, or ask for specific tasks necessary to complete the MAS-p (e.g., opening the mouth to assess post-swallow residuals in the oral cavity), but will not want to propose any additional requests nor can dietary instructions be given unless necessary for patient safety. No special/facilitative position will be asked. Each patient will be allowed to choose the food to eat, respecting any consistency constraints indicated by previous swallowing assessments. The assessment will be considered completed once the meal is finished. Each patient will be assessed at mealtime by two experienced speech therapists, informed of the protocol: scores obtained at MAS-p will be recorded independently and blinded to each other, to study inter-operator reliability. The assessment will be repeated after 48 hours, a time considered optimal in order to avoid possible bias related to the clinical improvement of the patient undergoing rehabilitation treatment, by one of the two speech therapists in order to study intra-operator reliability.

In group 3, i.e., those hospitalized patients who will be identified as suitable for diet modification during speech therapy, an endoscopic evaluation by videofluorographic swallowing study (VFSS), the gold standard for instrumental assessment of dysphagia, will be performed in advance by trained personnel before diet modification in order to verify that patients can tolerate a diet of different consistency; in this case, the observation of speech therapists during the meal and the completion of the MAS-p will be conducted both before (time 0) and after (time 1) the modification of the dietary pattern; thus the responsiveness of the scale will be assessed.

Regarding construct validity, the results of the scale will be compared with the results of two reliable and validated instruments for the assessment of dysphagia in pediatric settings, namely Montreal Children's Hospital Feeding Scale (MCH-FS) and Oral Motor Assessment Scale (OMAS), administered at the same time as the patient's first assessment by a speech therapist.

ELIGIBILITY:
Inclusion Criteria:

* Age between 24 months and 18 years
* Presence of risk factors for swallowing disorders of different etiology and severity at clinical evaluation
* Tolerance to exclusive oral feeding of a full or partial meal

Exclusion Criteria:

* Exclusive use of alternative feeding methods: nasogastric tube, percutaneous endoscopic gastrostomy (PEG), percutaneous endoscopic gastro-jejunal (PEG J)
* Absent or non-compliant caregiver

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This observational study examines subjects at risk for swallowing disorders. Subjects will be enrolled after clinical and speech evaluation in inpatient and outpatient settings.
  Competitive recruitment is planned among the involved centers IRCCS Fondazione Don Gnocchi ONLUS of Florence, Azienda Ospedaliero-Universitaria Meyer of Florence, Centro Bignamini Fondazione Don Gnocchi ONLUS of Falconara Marittima (AN), until the total of 240 subjects is reached.
  The signing of an informed consent to participate in the study by the subject's parent or legal guardian and compliance with the following inclusion and exclusion criteria is required.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Mealtime Assessment Scale - pediatric (MAS-p) adaptation | February - March 2022
  Drafting of the MAS-p scale as an adaptation of the MAS scale to the pediatric population 0 best value - 26 worst value
Meal Assessment Scale-pediatric (MAS-p) validation: internal consistency | March - August 2022
  Internal consistency is evaluated using Cronbach's alpha. In addition, Cronbach's alpha without an item was computed to identify whether the exclusion of the item would improve internal consistency. A good internal consistency is assumed in the presence of Cronbach's alpha > 0.70
Meal Assessment Scale-pediatric (MAS-p) validation: intra-rater agreement | March - August 2022
  The intra-rater agreement was evaluated by Intraclass Correlation Coefficient (ICC). An ICC above 0.75 was considered as indicating good agreement
Meal Assessment Scale-pediatric (MAS-p) validation: inter-rater agreement | March - August 2022
  Inter-rater agreement was tested using the average deviation index (AD index). A good inter-rater agreement was considered for an AD index below 0.66
Meal Assessment Scale-pediatric (MAS-p) validation: discriminative ability | March - August 2022
  The discrimination index was used to measure each item's ability to discriminate between those who scored high on the scale and those who scored low. The index was calculated for each item of the subscales Swallowing safety during the meal and Swallowing efficacy during the meal. The discrimination index was calculated as the difference between the number of individuals with a total score above the median who scored positive (2 or 3) on the item and the number of individuals with a total score below the median who scored positive on the item divided by the number of individuals above the median. Values above 0.4 were considered high, and above 0.2 desirable

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Cristella, MD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi Onlus, Florence, Italy

REFERENCES:
- [Background] Lawlor CM, Choi S. Diagnosis and Management of Pediatric Dysphagia: A Review. JAMA Otolaryngol Head Neck Surg. 2020 Feb 1;146(2):183-191. doi: 10.1001/jamaoto.2019.3622. PMID 31774493
- [Background] Bhattacharyya N. The prevalence of pediatric voice and swallowing problems in the United States. Laryngoscope. 2015 Mar;125(3):746-50. doi: 10.1002/lary.24931. Epub 2014 Sep 15. PMID 25220824
- [Background] Quitadamo P, Thapar N, Staiano A, Borrelli O. Gastrointestinal and nutritional problems in neurologically impaired children. Eur J Paediatr Neurol. 2016 Nov;20(6):810-815. doi: 10.1016/j.ejpn.2016.05.019. Epub 2016 Jun 11. PMID 27397730
- [Background] Arvedson JC. Assessment of pediatric dysphagia and feeding disorders: clinical and instrumental approaches. Dev Disabil Res Rev. 2008;14(2):118-27. doi: 10.1002/ddrr.17. PMID 18646015
- [Background] Rogers B, Arvedson J. Assessment of infant oral sensorimotor and swallowing function. Ment Retard Dev Disabil Res Rev. 2005;11(1):74-82. doi: 10.1002/mrdd.20055. PMID 15856438
- [Background] Majnemer A, Snider L. A comparison of developmental assessments of the newborn and young infant. Ment Retard Dev Disabil Res Rev. 2005;11(1):68-73. doi: 10.1002/mrdd.20052. PMID 15856441
- [Background] Barton C, Bickell M, Fucile S. Pediatric Oral Motor Feeding Assessments: A Systematic Review. Phys Occup Ther Pediatr. 2018 May;38(2):190-209. doi: 10.1080/01942638.2017.1290734. Epub 2017 Apr 21. PMID 28430014
- [Background] Ramsay M, Martel C, Porporino M, Zygmuntowicz C. The Montreal Children's Hospital Feeding Scale: A brief bilingual screening tool for identifying feeding problems. Paediatr Child Health. 2011 Mar;16(3):147-e17. doi: 10.1093/pch/16.3.147. PMID 22379377
- [Background] Ortega Ade O, Ciamponi AL, Mendes FM, Santos MT. Assessment scale of the oral motor performance of children and adolescents with neurological damages. J Oral Rehabil. 2009 Sep;36(9):653-9. doi: 10.1111/j.1365-2842.2009.01979.x. Epub 2009 Jul 15. PMID 19627455
- [Background] Sanchez K, Spittle AJ, Allinson L, Morgan A. Parent questionnaires measuring feeding disorders in preschool children: a systematic review. Dev Med Child Neurol. 2015 Sep;57(9):798-807. doi: 10.1111/dmcn.12748. Epub 2015 Mar 24. PMID 25809003
- [Background] Myer CM 4th, Howell RJ, Cohen AP, Willging JP, Ishman SL. A Systematic Review of Patient- or Proxy-Reported Validated Instruments Assessing Pediatric Dysphagia. Otolaryngol Head Neck Surg. 2016 May;154(5):817-23. doi: 10.1177/0194599816630531. Epub 2016 Apr 5. PMID 27048665
- [Background] Reilly S, Skuse D, Mathisen B, Wolke D. The objective rating of oral-motor functions during feeding. Dysphagia. 1995 Summer;10(3):177-91. doi: 10.1007/BF00260975. PMID 7614860
- [Background] Pizzorni N, Valentini D, Gilardone M, Borghi E, Corbo M, Schindler A. The Mealtime Assessment Scale (MAS): Part 1 - Development of a Scale for Meal Assessment. Folia Phoniatr Logop. 2020;72(3):169-181. doi: 10.1159/000494135. Epub 2019 Apr 18. PMID 30999311
- [Background] Pizzorni N, Valentini D, Gilardone M, Scarponi L, Tresoldi M, Barozzi S, Corbo M, Schindler A. The Mealtime Assessment Scale (MAS): Part 2 - Preliminary Psychometric Analysis. Folia Phoniatr Logop. 2020;72(3):182-193. doi: 10.1159/000494136. Epub 2019 Apr 17. PMID 30995652
- [Background] Hansen T, Lambert HC, Faber J. Reliability of the Danish version of the McGill Ingestive Skills Assessment for observation-based measures during meals. Scand J Occup Ther. 2012 Nov;19(6):488-96. doi: 10.3109/11038128.2012.674552. Epub 2012 May 1. PMID 22545775
- [Background] Ortega Ade O, Marques-Dias MJ, Santos MT, Castro T, Gallottini M. Oral motor assessment in individuals with Moebius syndrome. J Oral Pathol Med. 2014 Feb;43(2):157-61. doi: 10.1111/jop.12107. Epub 2013 Aug 10. PMID 23930941
- [Background] Kaviyani Baghbadorani M, Soleymani Z, Dadgar H, Salehi M. The effect of oral sensorimotor stimulations on feeding performance in children with spastic cerebral palsy. Acta Med Iran. 2014;52(12):899-904. PMID 25530052
- [Background] Arvedson JC, Lefton-Greif MA. Instrumental Assessment of Pediatric Dysphagia. Semin Speech Lang. 2017 Apr;38(2):135-146. doi: 10.1055/s-0037-1599111. Epub 2017 Mar 21. PMID 28324903